CLINICAL TRIAL: NCT04196205
Title: Study Evaluating the Safety and Efficacy With Anti-CD19 CAR-T Cells for Relapsed or Refractory Acute Lymphoblastic Leukemia and Lymphomas
Brief Title: Anti-CD19 CAR-T Cells for Relapsed or Refractory Acute Lymphoblastic Leukemia and Lymphomas
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, LiFei, M.D.,Ph.D., The First Affiliated Hospital of Nanchang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018027
Record Dates: First submitted 2019-12-09; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Acute Lymphoblastic Leukemia ,Lymphomas
Keywords: acute lymphoblastic leukemia ;Lymphomas

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anti-CD19 CAR-T (Experimental): Anti-CD19 CAR-T
  Interventions: Biological: Anti-CD19 CAR-T

INTERVENTIONS:
Biological: Anti-CD19 CAR-T — 1 - 2×10^6 Anti-CD19 CAR-T cells/kg body weigh

SUMMARY:
This is a single arm, open-label, single center study to determine the safety and efficacy of Anti-CD19 CAR-T cells in patients with relapsed or refractory acute lymphoblastic leukemia and Lymphomas.

DETAILED DESCRIPTION:
CD19 has been extensively evaluated as a therapeutic target for relapsed or refractory B cell malignancy by chimeric antigen receptor T cell therapy,this is a single arm, open-label, single center study to determine the safety and efficacy of Anti-CD19 CAR-T cells in patients with refractory acute lymphoblastic leukemia and Lymphomas.

ELIGIBILITY:
Inclusion Criteria: Subjects diagnosed as Relapsed or Refractory acute lymphoblastic leukemia and Lymphomas ，and have no effective treatment option (such as autograft or allogeneic stem cell transplantation) and estimated survival time of the current treatment < 2 years, The specific requirements are as follows:

1. Male or female aged 18-70 years old ;
2. Estimated Survival time > 12 weeks;
3. Relapsed and refractory acute lymphoblastic leukemia and lymphoma were confirmed by physical examination, pathological examination, laboratory examination and imaging;
4. Chemotherapy failure or recurrent acute lymphoblastic leukemia and Lymphomas;
5. Glutamic-pyruvic transaminase, glutamic oxalacetic transaminase< 3 fold of normal level;
6. Bilirubin<2.0mg/dl;
7. Karnofsky Performance Status>50% at the time of screening;
8. Adequate pulmonary, renal, hepatic, and cardiac function;
9. Fail in autologous or allogenic haemopoietic stem cell transplantation;
10. Not suitable for stem cell transplantation conditions or abandoned due to conditions;
11. Free of leukocytes removal contraindications;
12. Voluntarily join CAR-T clinical trial ,Understand and sign written informed consent.

Exclusion Criteria:

1. The patient is a pregnant or breastfeeding woman, or is a woman with a pregnancy plan within six months;
2. Patients have infectious diseases (such as HIV, active tuberculosis, etc.);
3. The patient is an active hepatitis B or hepatitis C infection;
4. Feasibility assessment proves that the efficiency of transduction of lymphocyte is below 10% or the lymphocyte cannot be propagated ;
5. Abnormal vital signs;
6. Subjects with mental or psychological illness who cannot be combined with treatment and efficacy evaluation;
7. Highly allergic constitution or history of severe allergies, especially allergy to interleukin-2;
8. General infection or local severe infection, or other infection that is not controlled;
9. Dysfunction in lung, heart, kidney and brain;
10. Severe autoimmune diseases;
11. Other symptoms that are not applicable for CAR-T.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-12-01 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall responce rate(ORR) | 2 years
  Assessment of ORR (ORR = CR+PR ) at 2 months of treatment
Overall survival (OS) | 2 years
  Assessment of OS(Overall survival) at 6 months of treatment
Progression-free survival (PFS) | 2 years
  Assessment of PFS(Progression-free survival ) at 6 months of treatment
minimal residual disease（MRD） | 2 years
  Assessment of MRD negative overall response rate at 3 months of treatment

SECONDARY OUTCOMES:
Safety (incidence of adverse events defined as dose-limited toxicity) | Study treatment until Week 24
  Occurrence of study related adverse events defined as NCI CTCAE 4.0 > grade 3 possibly, probably, or definitely related to study treatment.
Expression of CD19 CART cells | 2 years
  Expression of CD19 CART cells detected by flow cytometry in blood and bone marrow.
Detection of CD19 CART cells | 2 years
  Detection of CD19 CART cells in blood, bone marrow by Quantitative Polymerase Chain Reaction (q-PCR).

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nangchang University, Nanchang, Jiangxi, China